CLINICAL TRIAL: NCT05114044
Title: The Effects of Core Stability Training on Functional Ability and Muscle Thickness in Chronic Stroke Patients
Brief Title: The Effects of Core Stability Training in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Sefa Gümrük Aslan, Consultant Physiatrist, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23
Record Dates: First submitted 2021-10-20; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core stability group (Experimental): Patients were performed therapy 5 times a week for 45 min over a period of 3 weeks. The therapy session takes 45 min; 15 min of the session was core stability training, remaining 30 min were conventional therapy.
  Interventions: Other: Core stability training
- Conventional therapy group (Active Comparator): Patients were performed therapy 5 times a week for 45 min over a period of 3 weeks. The therapy session takes 45 min of conventional therapy.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: Core stability training — The core stability training were performed 5 days a week for 15 min over a period of 3 weeks. The conventional therapy were performed 5 days a week for 30 min (remaining time of each session) over a period of 3 weeks. Duration of each session was 45 min.
  Arms: Core stability group
Other: Conventional therapy — The conventional therapy were performed 5 days a week for 45 min over a period of 3 weeks. Duration of each session was 45 min
  Arms: Conventional therapy group

SUMMARY:
The purpose of this study is to assess effects of core stability training on functional ability, balance, gait, motor functions, quality of lite and core muscle thickness of chronic stroke patients.

DETAILED DESCRIPTION:
After being informed about the study all the patients giving written informed consent were assessed. At the beginning the eligible patients were randomized into two groups: core stability and conventional therapy group. The therapy programs were performed 5 times a week for 45 min over a period of 3 weeks. Patients were assessed twice: before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* First onset
* Stroke duration from 6 months to 2 years
* With ability to cooperate
* Independent ambulation or ambulation with assistive device

Exclusion Criteria:

* Uncooperative
* Neglect syndrome
* Surgical history of abdominal and hip region
* Drugs that affect neuromuscular control
* Other neurological disorders
* Serious diseases, unstable medical condition
* BMI ≥ 35

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline score of Berg Balance Scale at week 3 | Baseline and week 3 (after treatment)
  Berg Balance Scale is reliable and valid tool to assess balance and functional mobility. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function.
Change from baseline score of Motricity Index Scale for lower extremity at week 3 | Baseline and week 3 (after treatment)
  The Motricity Index was used to measure strength in upper and lower extremities after stroke. Assessing lower extremity strength is a 3 item list with each item consisting of a six point scale ranging from 0 to 33 (0, 9, 14, 19, 25, 33).
Change from baseline score of Trunk Control Test at week 3 | Baseline and week 3 (after treatment)
  Trunk Control Test assess four simple aspect of trunk movement. Total score range: 0 to 100.
Change from baseline score of 6 Minute Walk Test (6MWT) at week 3 | Baseline and week 3 (after treatment)
  6MWT is valid and reliable test to assess walking capacity of stroke patients. The distance that a patient can walk within six minutes is evaluated.
Change from baseline score of Functional Independence Measure (FIM) at week 3 | Baseline and week 3 (after treatment)
  FIM is valid and reliable scale to assess and grade the functional status of a person based on the level of assistance he or she requires. FIM is an 18-item, seven-level, ordinal scale intended to be sensitive to changes over the course of a comprehensive inpatient medical rehabilitation program.
Change from baseline score of Trunk Impairment Scale (TIS) at week 3 | Baseline and week 3 (after treatment)
  TIS is a tool to assess static and dynamic sitting balance and trunk coordination in a sitting position. On the static and dynamic sitting balance and coordination subscales the maximal scores that can be attained are 7, 10 and 6 points.
Change from baseline score of Timed Up and Go Test (TUG) at week 3 | Baseline and week 3 (after treatment)
  TUG test is an assessment tool for measuring mobility in stroke patients. The TUG times a patient standing from a chair, walking 3 metres and returning to sit down.
Change from baseline score of Stroke Specific Quality of Life Scale (SS-QOL) at week 3 | Baseline and week 3 (after treatment)
  SS-QOL is a patient-centered outcome measure intended to provide an assessment of health-related quality of life specific to patients with stroke. Patients must respond to each question of the SS-QOL with reference to the past week. It is a self-report scale containing 49 items. Items are rated on a 5-point Likert scale.
Change from baseline measurements Core muscle thickness at week 3 | Baseline and week 3 (after treatment)
  Thickness of five core muscles (rectus abdominis, external oblique, internal oblique, transversus abdominis, multifidus and gluteus medius) are measured by ultrasound. Paretic and nonparetic side of each patient are assessed twice (at baseline and after treatment).

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)